CLINICAL TRIAL: NCT02108795
Title: The Effect of Remifentanil Infusion During Emergence on the Incidence of Emergence Delirium After Sevoflurane Anesthesia in Pediatric Strabismus Surgery
Brief Title: The Effect of Remifentanil Infusion During Emergence on the Incidence of Emergence Delirium
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yeungnam University College of Medicine (Other)
Responsible Party: Principal Investigator, Sangjin Park, assistant professor, Yeungnam University College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: apsj20140331
Record Dates: First submitted 2014-03-31; First posted 2014-04-09 (Estimated); Last update posted 2015-07-16 (Estimated); Status verified 2015-07

CONDITIONS: Delirium
MeSH Terms: conditions — Delirium | interventions — Remifentanil

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- remifentanil group (Experimental): Remifentanil 0.05 ug/kg/min is infused to the patients.
  Interventions: Drug: Remifentanil
- control (Placebo Comparator): Normal saline 0.2 ml/kg/hour is infused to the patients
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Remifentanil — Children randomised to remifentanil group receive remifentanil 0.05 ug/kg/min. Children randomised to control group receive normal saline (placebo)
  Other Names: remifentanil (ultiva)
  Arms: remifentanil group
Drug: Placebo
  Arms: control

SUMMARY:
The aim of the present study is to assess the effect of postoperative remifentanil infusion on the incidence of emergence agitation in preschool-aged children undergoing strabismus surgery with sevoflurane anaesthesia.

DETAILED DESCRIPTION:
Patients are randomly assigned to one of two groups. Anesthesia is maintained with sevoflurane and remifentanil infusion. All patients received a predetermined concentrations of remifentanil according to their group assignments (control group, remifentanil 0 ug/kg/min; remifentanil group, remifentanil 0.05 ug/kg/min) from 10 minutes before the end of surgery to discharge from postanesthetic care unit. emergence agitation is assessed during the emergence phase.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical status I and II
* preschool-aged children undergoing strabismus surgery

Exclusion Criteria:

* psychological disorders
* emotional disorders
* abnormal cognitive development
* developmental delay
* allergy to the drugs in our protocol

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 86 (Estimated)
Dates: Start 2014-04; Primary Completion 2016-04 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
the scale of emergence agitation | up to 30 minutes after arrival in postanesthetic care unit, and 30 minutes after discharge from postanesthetic care unit.
  A blinded observer record emergence agitation at just after laryngeal mask removal, 5 minutes after arrival in postanesthetic care unit, 10 minutes after arrival in postanesthetic care unit, 15 minutes after arrival in postanesthetic care unit, 30 minutes after arrival in postanesthetic care unit, and 30 minutes after discharge from postanesthetic care unit.

SECONDARY OUTCOMES:
the effect of remifentanil on the emergence | up to 30 minutes after the discharge form postanesthetic care unit
  A blinded observer record duration of anaesthesia, eye-opening time, time to remove laryngeal mask airway, respiratory depression, nausea, and vomiting at the end of surgery, 5 minutes after arrival in postanesthetic care unit, 10 minutes after arrival in postanesthetic care unit, 15 minutes after arrival in postanesthetic care unit, 30 minutes after arrival in postanesthetic care unit, and 30 minutes after discharge from postanesthetic care unit.

CONTACTS AND LOCATIONS:
Overall Officials: Sangjin Park, M.D., Principal Investigator — Department of Anesthesiology and Pain Medicine, College of medicine, Yeungnam University, Daemyung-Dong, Nam-Gu, Daegu, Republic of Korea
Locations (1):
- Department of Anesthesiology and Pain Medicine, Yeungnam University hospital, Daegu, South Korea